CLINICAL TRIAL: NCT06505252
Title: Comparison of Topical Use of Platelet-rich Plasma Versus Hyaluronic Acid During Endoscopic Fat Graft Myringoplasty
Brief Title: Comparison of Topical Use of Platelet-rich Plasma Versus Hyaluronic Acid During Endoscopic Fat Graft Myringoplasty: a Randomized Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Abdel-Hameed, assistant lecture of otolaryngeology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Endoscopic fat Myringoplasty
Record Dates: First submitted 2024-07-03; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Chronic Suppurative Otitis Media
Keywords: CSOM; chronic suppurative otitis media; tympanic membrane perforation; TM perforation; myringoplasty; tympanoplasty; endoscopic tympanoplasty
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to two groups:
  By using an online research randomizer (http://www.randomizer.org), patients will be randomly allocated to two groups Group (A): will do endoscopic myringoplasty using fat graft augmented by hylourinic acid Group (B): will do endoscopic myringoplasty using fat graft with PRP
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA group or group A (Experimental): * All patients underwent operations under general anesthesia. A single surgeon will perform all surgeries.
  * A small incision in the rim of ear lobule on the same side of the operated ear, a small piece of adipose tissue will be removed according to the experience of the surgeon.
  * The incision will be closed with vicryl 4/0 sutures.
  * Using 0 angulation endoscope visualization, the edges of the perforation will be refreshed and deepithelialized with a sharp Rosen's needle or sickle knife.
  * sponge gel (Gelfoam) will pushed through TM perforation into the middle ear to support the graft and to avoid its medialization. The previously removed fat graft will be inserted through the perforation adjusted so most of the fat piece lying medial to the perforation and small part laterally. HA was used in liquid form, using a 2 mL vial (® Hyalgan) containing 20 mg of sodium hyaluronate that is synthesized by fermentation. The vial will be prepared for direct injection.
  Interventions: Procedure: enoscopic Myringoplasty
- PRP group or group B (Experimental): * All patients underwent operations under general anesthesia. A single surgeon will perform all surgeries.
  * A small incision in the rim of ear lobule on the same side of the operated ear, a small piece of adipose tissue will be removed according to the experience of the surgeon.
  * The incision will be closed with vicryl 4/0 sutures.
  * Using 0 angulation endoscope visualization, the edges of the perforation will be refreshed and deepithelialized with a sharp Rosen's needle or sickle knife.
  * sponge gel (Gelfoam) will pushed through TM perforation into the middle ear to support the graft and to avoid its medialization The previously removed fat graft will be inserted through the perforation adjusted so most of the fat piece lying medial to the perforation and small part laterally PRPG was inserted into the external auditory canal (EAC) on the outer face of the TM remnant and fat graft. Special attention will be given to obtaining close contact among the PRPG, TM, and fat graft. The
  Interventions: Procedure: enoscopic Myringoplasty

INTERVENTIONS:
Procedure: enoscopic Myringoplasty — general anesthesia. A single surgeon will perform all surgeries.
  * A small incision in the rim of ear lobule on the same side of the operated ear, a small piece of adipose tissue will be removed according to the experience of the surgeon.
  * Using 0 angulation endoscope visualization, the edges of the perforation will be refreshed and deepithelialized with a sharp Rosen's needle
  * sponge gel (Gelfoam) will pushed through TM perforation into the middle ear to support the graft and to avoid its medialization
  * the previously removed fat graft will be inserted through the perforation adjusted so most of the fat piece lying medial to the perforation and small part laterally in patients group A: 0.5 mL of HA vial will be injected directly over the fat graft and the TM remnant. After 5 minutes small gelfoam pieces soaked in 0.5 mL of HA vial will applied over the fat in patients group B PRPG was inserted into the external auditory canal on the outer face of the TM remnant and fat

SUMMARY:
This study aimed to compare the effect of adding HA versus PRP to endoscopic FGM in cases of small or medium-sized central TM perforation in the form of:

1. Evaluation of the graft uptake rate.
2. Evaluation and comparing audiological outcomes.
3. Finding out intraoperative and postoperative morbidity.

DETAILED DESCRIPTION:
Tympanic membrane (TM) perforations result in recurrent middle ear infection and hearing loss. Both these hazards can be prevented by the reconstructive surgery of the tympanic membrane.

Fat graft myringoplasty (FGM) has been reported as a suitable procedure to close long-standing TM perforations FGM is an efficient, safe and potentially fast method for TM perforation repairing with a success rate varies from 79% to 91%..Many researches was done to use supporting material in myringoplasty Saliba et al used hyaluronic acid fat graft myringoplasty [HAFGM] and results in a higher success rate than using FGM alone. El-Anwar et al proved that Topical autologous platelet-rich plasma(PRP) application during myringolpasty is safe, efficient and enhances healing of TM perforation PRP includes many autologous growth factors that have significant functions like cell proliferation, migration, and angiogenesis. Fibrin and fibronectin are essential proteins in PRP that provide the structural support needed for the cell migration, cell proliferation, and 3-dimensional growth of tissues.

HA has been shown to play a role in cellular signaling, leukocyte growth and migration, Cell adhesion and biological remodeling and is mainly involved in tissue healing with a central role in modulating inflammatory responses also, Its absorption of water causes expansion in volume and formation of a viscoelastic gel which constitutes a favorable scaffold for tissue regeneration and remodeling .

ELIGIBILITY:
Inclusion Criteria:

* Patients with central small or median sized dry perforation
* Aged between 14 and 50 years
* In cases of CSOM the perforation must be dry with no otorrhea with healthy middle ear mucosa for at least three month without medications
* Conductive gap on audiometry not more than 40 dB.

Exclusion Criteria:

* Discharging CSOM .
* Concurrent URTI .
* CSOM with dry marginal perforation
* Patients who didn't come for follow up.
* Age less than 14 or more than 50.
* Unsafe CSOM with cholesteatoma, apparent retraction pockets, granulations, or extensive myringosclerosis reaching the edges of the perforation. Patients
* Patients who are suspected of having Eustachian tube dysfunction.
* Suspected ossicular pathology in safe CSOM if the ABG > 40dB.
* Patients with history of Previous ear surgery.
* Patients unfit for surgery or having chronic medical illness.
* Narrow external auditory canal.
* Patients who refused to enrolled in our study
* Patients with sensorineural hearing loss or only functioning ear.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
graft taking | 3 months
  Endoscopic examination of TM: Graft will considered as successfully taken if there is no residual TM perforation after 3 months postoperativly.

SECONDARY OUTCOMES:
Audiotympanogram | 3 months
  effect on hearing by using Audiotympanogram will be done three months post-operative
Otorrhea | 1 month
  presence or absence of otorrhea by history and ear examination

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Anwar MW, El-Ahl MA, Zidan AA, Yacoup MA. Topical use of autologous platelet rich plasma in myringoplasty. Auris Nasus Larynx. 2015 Oct;42(5):365-8. doi: 10.1016/j.anl.2015.02.016. Epub 2015 Mar 17. PMID 25794691
- [Background] Knutsson J, Kahlin A, von Unge M. Clinical and audiological short-term and long-term outcomes of fat graft myringoplasty. Acta Otolaryngol. 2017 Sep;137(9):940-944. doi: 10.1080/00016489.2017.1326063. Epub 2017 May 24. PMID 28537107
- [Background] Kim HC, Park KS, Yang HC, Jang CH. Surgical results and factors affecting outcome in patients with fat-graft myringoplasty. Ear Nose Throat J. 2024 Jul;103(7):442-446. doi: 10.1177/01455613211063243. Epub 2021 Dec 9. PMID 34881650